CLINICAL TRIAL: NCT05223166
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Clinical Study to Evaluate the Efficacy and Safety of Pitolisant in the Treatment of Excessive Daytime Sleepiness in Patients With Obstructive Sleep Apnea
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of Pitolisant in the Treatment of EDS in Patients With OSA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Citrine Medicine Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSPIT32101
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Excessive Daytime Sleepiness
MeSH Terms: conditions — Disorders of Excessive Somnolence | interventions — pitolisant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pitolisant (Experimental): Histamine H3 receptor H3R antagonist/ inverse agonist
  Interventions: Drug: Pitolisant
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Pitolisant — Wakix tablet
  Arms: Pitolisant
Drug: Placebo oral tablet — Matching placebo tablets will be provided for each strength of active pitolisant film-coated tablets.
  Arms: Placebo

SUMMARY:
The objective of this study is to demonstrate the efficacy and safety of pitolisant versus placebo during 12 weeks of the Double Blind period, to treat the Excessive Daytime Sleepiness (EDS) in patients with Obstructive Sleep Apnea (OSA) not tolerating or refusing the nasal Continuous Positive Airway Pressure (nCPAP) therapy or treated by nCPAP but still complaining of EDS.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria

  1. Voluntarily participate in the clinical study; fully understand and know the study and sign the informed consent form (ICF); willing to follow and able to complete all study procedures;
  2. Male or female aged 18 years to 70 years;
  3. Subjects affected by Obstructive Sleep Apnoea (OSA) with excessive daytime sleepiness;
  4. Female subjects of childbearing potential must have a negative serum pregnancy test 1 week before the first dose; female subjects or male subjects with a spouse of childbearing potential must agree to take contraceptive measures from the signing of the informed consent form to 1 months after the last dose of study drug;
  5. Subjects must be willing not to operate a car (if sleepy at wheel) or heavy machinery for the duration of the study or as long as the investigator deems it clinically indicated. In addition, subjects need to be willing to maintain daily behaviors (e.g., circadian rhythm, caffeine intake, nocturnal sleep duration, etc.) during the study that may affect their daytime sleepiness.

Exclusion Criteria:

1. Participated in any other drug clinical trial or receiving other clinical trial treatment within 30 days before the first dose;
2. Subjects who have previously received pitolisant, either from other clinical studies of pitolisant or from the subject use program, or from treatment with commercially available pitolisant (Wakix ®);
3. Use of prohibited drugs specified in the protocol within 14 days before enrollment;
4. The mean oxygen saturation < 85% or the lowest oxygen saturation < 70% by PSG.
5. Acute or chronic diseases affecting efficacy evaluation, such as severe chronic obstructive pulmonary disease (COPD);
6. Previous history of drug, alcohol, narcotic or other drug abuse or dependence;
7. Any serious cardiovascular system abnormalities (e.g., ischemic cardio-cerebral disease), such as recent myocardial infarction, angina, severe hypertension or arrhythmia in the recent 6 months, ECG Fridericia-corrected QT interval higher than 450 ms, history of left ventricular hypertrophy or mitral valve prolapse;
8. Subjects with severe co-morbid medical or biological conditions that may jeopardize participation in the study (especially cardiovascular system problems and unstable diabetes) as judged by the investigator;
9. Any positive serology test for HIV, HCV, HBsAg and syphilis;
10. Female subjects who are pregnant or breast-feeding;
11. Known or suspected hypersensitivity to study drug or to any excipients;
12. Cognitive impairment due to any psychiatric or neurological condition, including epilepsy and dementia, which may limit the understanding, execution of the informed consent form, and compliance of the study;
13. Presence of severe hepatic insufficiency (Child Pugh C) or severe renal impairment (eGFR<30 ml/min/1.73㎡), or other significant abnormalities in physical examination/clinical laboratory tests, and any clinically significant condition that may interfere with the subject's completion of the study;
14. Subjects who are judged by the investigator to be unsuitable for this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline of ESS | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tsinghua Changgung Hospital, Beijing, China